CLINICAL TRIAL: NCT00564564
Title: Quetiapine Augmentation Versus Clomipramine Augmentation of Selective Serotonin Reuptake Inhibitors for Obsessive-compulsive Disorder Patients That do Not Respond to a SSRI Trial: a Randomized Open-trial.
Brief Title: Quetiapine Augmentation Versus Clomipramine Augmentation of SSRI for Obsessive-compulsive Disorder Patients
Acronym: QCAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Juliana Belo Diniz, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 968/05; 2005/55628-08 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Obsessive Compulsive Disorder
Keywords: obsessive compulsive disorder; pharmacological treatment; quetiapine; clomipramine; SSRI
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Quetiapine Fumarate; Clomipramine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quetiapine augmentation (Experimental): Quetiapine up to 200mg/day plus SSRI at maximum tolerated or recommended dosage
  Interventions: Drug: Quetiapine
- Clomipramine augmentation (Active Comparator): Clomipramine up to 150mg/day plus SSRI at maximum tolerated or recommended dosage
  Interventions: Drug: Clomipramine

INTERVENTIONS:
Drug: Quetiapine — Quetiapine once a day at maximum dosage of 200mg per day asociated to a SSRI (maximum dosage of 40mg per day for fluoxetine; 200mg per day for sertraline and 60mg per day for citalopram)
  Other Names: Seroquel
  Arms: Quetiapine augmentation
Drug: Clomipramine — Clomipramine once a day at maximum dosage of 75mg per day plus SSRI (maximum dosage of 40mg per day for fluoxetine; 200mg per day for sertraline and 60mg per day for citalopram)
  Other Names: Anafranil
  Arms: Clomipramine augmentation

SUMMARY:
The objective of this trial is to compare in an open trial format the efficacy of association of clomipramine and quetiapine with SSRI after SSRI treatment failed to produce complete remission of obsessive compulsive disorder symptoms.

DETAILED DESCRIPTION:
The objective of this trial wis to compare in an randomized open trial format the efficacy of association of clomipramine at maximum dosage of 75mg per day and quetiapine at maximum dosage of 200mg per day with SSRI after SSRI treatment for 12 weeks failed to produce complete remission of OCD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* primary OCD diagnosis according to DSM IV criteria
* current symptoms were responsible for significant distress
* previous trial of at least 12 weeks with SSRI (being at least 8 weeks at maximum tolerated dosage) failed to produce full remission of OCD symptoms

Exclusion Criteria:

* presence of clinical or neurological diseases that may be worsen by the medications included in treatment protocol
* current substance dependence or abuse,
* current psychotic symptoms
* current suicide risk
* and current pregnancy or intention to get pregnant before the end of the treatment protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
YBOCS | 12 weeks
  difference between initial and final (12 week) Yale Brown Obsessive Compulsive Scale (YBOCS)score

SECONDARY OUTCOMES:
CGI | 12 weeks
  Clinical Global Impression score for improvement at week 12
Tolerability | weeks 0,2,4,8 and 12
  adverse events measure (emphasis in serotonergic syndrome)
Cardiotoxicity | week 0 and 2
  Changes in baseline (week 0) EKG regarding QT interval

CONTACTS AND LOCATIONS:
Overall Officials: Juliana B Diniz, MD, Principal Investigator — Department of Psychiatry University of São Paulo Medical School
Locations (1):
- Institute of Psychiatry, Clinics Hospital, University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Bloch MH, Landeros-Weisenberger A, Kelmendi B, Coric V, Bracken MB, Leckman JF. A systematic review: antipsychotic augmentation with treatment refractory obsessive-compulsive disorder. Mol Psychiatry. 2006 Jul;11(7):622-32. doi: 10.1038/sj.mp.4001823. Epub 2006 Apr 4. PMID 16585942
- [Background] Browne M, Horn E, Jones TT. The benefits of clomipramine-fluoxetine combination in obsessive compulsive disorder. Can J Psychiatry. 1993 May;38(4):242-3. doi: 10.1177/070674379303800402. PMID 8518974
- [Background] Denys D, de Geus F, van Megen HJ, Westenberg HG. A double-blind, randomized, placebo-controlled trial of quetiapine addition in patients with obsessive-compulsive disorder refractory to serotonin reuptake inhibitors. J Clin Psychiatry. 2004 Aug;65(8):1040-8. doi: 10.4088/jcp.v65n0803. PMID 15323587
- [Background] Fineberg NA, Sivakumaran T, Roberts A, Gale T. Adding quetiapine to SRI in treatment-resistant obsessive-compulsive disorder: a randomized controlled treatment study. Int Clin Psychopharmacol. 2005 Jul;20(4):223-6. doi: 10.1097/00004850-200507000-00005. PMID 15933483
- [Background] Pallanti S, Quercioli L, Paiva RS, Koran LM. Citalopram for treatment-resistant obsessive-compulsive disorder. Eur Psychiatry. 1999 Apr;14(2):101-6. doi: 10.1016/s0924-9338(99)80725-1. PMID 10572334
- See also: institutional site — http://www.ipqhc.org.br/
- See also: Mains results — https://www.ncbi.nlm.nih.gov/pubmed/19164490